CLINICAL TRIAL: NCT04618835
Title: Exertional Desaturation as a Marker of Risk - Validation Study for the 40-steps-test; A Multi-centre Prospective Observational Cohort Study
Brief Title: Physical Activity a Vital Sign? 40 Steps to Safety Test for Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Betsi Cadwaladr University Health Board (Other Government)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr Christian P Subbe, Consultant Physician, Betsi Cadwaladr University Health Board
Other Study IDs: 283998
Record Dates: First submitted 2020-10-31; First posted 2020-11-06 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Medical Emergencies
Keywords: Exercise tolerance test; Vital signs; Readmission; Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency presentations: Patients discharged after a presentation to practitioners in the community, primary and secondary care.
  Interventions: Diagnostic Test: 40-Steps-test

INTERVENTIONS:
Diagnostic Test: 40-Steps-test — 40 steps performed on the spot

SUMMARY:
Exertional desaturation is a feature of COVID-19. The study will measure vital signs of patients discharge by practitioners in primary care, secondary care or by paramedic practitioners. Patients will then undertake a 40-steps on the spot walk followed by measurements of heart rate and oxygen saturations for up to two minutes. Association of desaturation with 30 days hospital admission and mortality will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients are being considered for discharge to independent care
* Participant is willing and able to give informed consent for participation in the study.
* Patient with independent, stable, gait
* Patient is alert, attentive, coherent, and calm
* Male or Female, aged 18 years or above.

Exclusion Criteria:

* Minor injuries
* Elective surgery patients
* Post-operative patients at discharge
* Requires supplemental oxygen
* Shortness of breath at rest (i.e. Borg or Numerical Rating Scale >=2)
* Unstable angina
* Patients on long-term-oxygen therapy
* Pregnancy as stated by patient
* Oxygen saturations < 95% on room air
* Resting heart rate > 100 bpm
* Resting respiratory rate > 25 bpm
* ECG with signs of acute ischemia in patients where an ECG has been requested by the treating clinician
* National Early Warning Score of 5 or more
* Nursing home residents, or those being transferred to a nursing home or similar care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All alert and mobile acutely ill patients with mild symptoms and little or no vital sign derangement being considered for discharge to independent care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-11-03 (Estimated); Study Completion 2021-11-03 (Estimated)

PRIMARY OUTCOMES:
Change in decision to discharge | 24 hours
  1. No change
  2. Further investigations
  3. Hospital admission
  a) No change b) Further investigations c) Hospital admission
Hospital | 30 days
  Admission to hospital within 30 days of the test
Death | 30 days
  Death within 30 days of the test

SECONDARY OUTCOMES:
Feasibility of the 40-steps test | 12 months
  Proportion of sites and patients able to undertake the test
Change in heart rate | Within 2 minutes of completion of the test
  Change in heart rate compared to value measured before expercise
Change in oxygen saturations | Within 2 minutes of completion of the test
  Change in heart rate compared to value measured before exercise
Change in respiratory rate | Within 2 minutes of completion of the test
  Change in respiratory rate compared to value measured before exercise
Change in breathlessness | Within 2 minutes of completion of the test
  Change in breathlessness compared to value measured before exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Ysbyty Gwynedd, Menai Bridge, Gwynedd, United Kingdom

IPD SHARING:
Plan to Share IPD: No